CLINICAL TRIAL: NCT05273905
Title: Augmented Velocity Index of Intra-abdominal, Carotid and Retinal Arteries: In Relation to Arterial Stiffness and Cardiovascular Risk Factors.
Brief Title: Augmented Velocity Index of Intra-abdominal, Carotid and Retinal Arteries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Liu Kin Hung, Adjunct Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2022.3.1
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Arterial Stiffness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound derived Avi — Assess the Avi of carotid arteries, hepatic arteries, renal arteries and central retinal arteries.

SUMMARY:
Background:

Augmented Velocity Index (Avi) is a new Doppler index which can potentially be used to assess arterial stiffness. The Avi of common carotid artery is found to be associated with arterial stiffness and have initial correlation with cardiovascular risk factors. Avi can be used in any vessels (superficial or deep vessels) where arterial Doppler waveforms can be obtained.

Aims:

The aims of this study are to investigate the associations of Avi of hepatic artery, renal artery, central retinal artery and internal carotid artery with arterial stiffness and cardiovascular risk factors in a group of apparently normal subjects.

Methods:

Recruit 350 subjects with no known medical illness or drug treatment for ultrasound examinations and blood tests. In ultrasound examination, the Avi of carotid arteries, hepatic arteries, renal arteries and retinal arteries are recorded. The carotid-femoral pulse wave velocity is also calculated for the assessment of central aortic stiffness.

Other important correlates of arterial stiffness including carotid intima-media thickness, fatty liver status, liver stiffness and abdominal fat thickness are assessed in the ultrasound examination.

The clinical and laboratory examinations include anthropometric indexes, plasma glucose level, lipid profile, renal function tests, liver function test, urinary albumin creatinine ratio, blood pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy volunteers

Exclusion Criteria:

* Subjects with known medical illnesses including cancer, stroke, cardiovascular disease, diabetes, hypertension, dyslipidaemia, peripheral vascular disease, gout, systemic lupus erythematosus, psoriasis, rheumatoid arthritis and thyrotoxicosis.
* Subjects with long term drug use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Augmented Velocity Index (Avi) | Aug 2022 - May 2024
  Avi of carotid, renal, hepatic and retinal arteries as recorded from the Doppler ultrasound waveforms of those arteries

SECONDARY OUTCOMES:
Arterial wall thickness, liver stiffness and fatty liver status | Aug 2022 - May 2024
  Intima-media thickness of carotid artery is measured in gray scale ultrasound images; Liver stiffness is assessed by shear wave elastography of ultrasound technique; Fatty liver status is determined by the attenuation imaging of ultrasound

IPD SHARING:
Plan to Share IPD: No